CLINICAL TRIAL: NCT00102414
Title: A Randomized Phase III Study Comparing Gemcitabine Plus Carboplatin Versus Carboplatin Monotherapy in Patients With Advanced Epithelial Ovarian Carcinoma Who Failed First-Line Platinum-Based Therapy
Brief Title: Gemcitabine Plus Carboplatin Versus Carboplatin Monotherapy in Patients With Advanced Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AGO Study Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR 2.5
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Last update posted 2006-11-14 (Estimated); Status verified 2005-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Recurrence or progression; Gemcitabine plus Carboplatin vs Carboplatin
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence; Disease Progression | interventions — Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine

SUMMARY:
The primary objective of this study is to compare the time to progressive disease in patients treated with gemcitabine plus carboplatin versus carboplatin monotherapy. Patients will have advanced epithelial ovarian cancer and have failed first-line platinum-containing therapy 6 months after treatment discontinuation.

DETAILED DESCRIPTION:
Carboplatin is commonly used for the treatment of ovarian cancer in first- and second-line therapy. The efficacy of gemcitabine in ovarian carcinoma was researched in various Phase 2 studies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven ovarian cancer with evidence of recurrence or progression
* Failed first-line platinum containing therapy after 6 months of treatment discontinuation
* Documented lesion as evidenced by appropriate computerized tomography (CT), magnetic resonance imaging (MRI) scan, chest x-ray, or ultrasound.
* Previous hormonal therapy or radiotherapy must be terminated at least 3 weeks before study drug administration
* Adequate bone marrow reserve: neutrophils ≥ 1.5 x 10^9/L and platelets ≥ 100 x 10^9/L

Exclusion Criteria:

* Receiving concomitant cytotoxic or other antineoplastic treatment. Hormone replacement therapy is allowed, as are steroid antiemetics
* Clinical evidence of central nervous system metastases
* Active infection
* Cannot adequately be followed up for the duration of the study
* A second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin)
* Use of any investigational agent in the 3 weeks prior to inclusion
* Serious concomitant systematic disorders incompatible with the study
* Received more than one previous chemotherapy regimen or had prior gemcitabine treatment
* Patients with tumor of borderline malignancy
* Patients with estimated GFR ≤ 50 mL/min

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356
Dates: Start 1999-09; Study Completion 2004-11

PRIMARY OUTCOMES:
Time to progressive disease

SECONDARY OUTCOMES:
Response rate
Duration of response
Survival time
Toxicity
Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Jacobus Pfisterer, Prof. Dr. med., Principal Investigator — AGO Study Group

REFERENCES:
- [Result] Pfisterer J, Plante M, Vergote I, du Bois A, Hirte H, Lacave AJ, Wagner U, Stahle A, Stuart G, Kimmig R, Olbricht S, Le T, Emerich J, Kuhn W, Bentley J, Jackisch C, Luck HJ, Rochon J, Zimmermann AH, Eisenhauer E; AGO-OVAR; NCIC CTG; EORTC GCG. Gemcitabine plus carboplatin compared with carboplatin in patients with platinum-sensitive recurrent ovarian cancer: an intergroup trial of the AGO-OVAR, the NCIC CTG, and the EORTC GCG. J Clin Oncol. 2006 Oct 10;24(29):4699-707. doi: 10.1200/JCO.2006.06.0913. Epub 2006 Sep 11. PMID 16966687